CLINICAL TRIAL: NCT07123571
Title: A Pilot Randomized Trial: Effectiveness of a Five-day Online Audio-visual Contagious Laughter Intervention to Enhance Well-being in Adults
Brief Title: A Five-Day Contagious Laughter Intervention for Adult Well-being
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zayed University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Laughter & Wellbeing
Record Dates: First submitted 2025-07-31; First posted 2025-08-14 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Well-being
Keywords: Well-being; Laughter
MeSH Terms: conditions — Laughter

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Contagious Laughter Intervention (Experimental)
  Interventions: Behavioral: Contagious Laughter
- Control (No Intervention): Control group without intervention

INTERVENTIONS:
Behavioral: Contagious Laughter — Contagious laughter videos
  Arms: Contagious Laughter Intervention

SUMMARY:
The goal of this pilot trial is to determine the effectiveness of a five day contagious laughter intervention on adult well-being. The main questions it aims to answer are:

Does exposure to a five-day online contagious laughter intervention improve subjective well-being in adults compared to waitlist controls? Does exposure to a five-day online contagious laughter intervention improve subjective mood status in adults compared to waitlist controls?

Participants in the intervention group will:

View a one-minute contagious laughter video each day for five days Complete the WHO5 Wellbeing index pre and post intervention Rate their mood status before and after each laughter video on each day of the intervention After viewing each video, rate how much they laughter along with the video on each day of the intervention

Participants in the waitlist control group will:

Complete the WHO5 wellbeing index at baseline and again after six days

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Resident of the United Arab Emirates
* Fluent in English and/or Arabic
* Access to a stable internet connection
* Access to a smartphone and/or laptop/tablet

Exclusion criteria:

* Children (<18 years old)
* Adults above 60 years old
* Those with cognitive and/or physical disabilities
* Those with hearing and/or vision impairment
* Illiterate, and/or individuals who did not (or were unable to) provide consent.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2022-09-15 (Actual); Primary Completion 2023-05-14 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Well-being | Well-being will be assessed at baseline (start of study) and will be reassessed on day six (one day after the five-day intervention). The final score range is 0-100 where 0 represents the worse possible well-being and 100 represents the best.
  Adult well-being will be assessed using the WHO5 Wellbeing Index (WBI)
  The WHO5 WBI is scored by summing the responses to five questions, each using a 6-point Likert scale (0-5). This derives a raw score between 0 and 25. This raw score is then multiplied by 4 to calculate a percentage score with a range of 0-100, where 0 represents the worst possible well-being and 100 represents the best.

SECONDARY OUTCOMES:
Subjective mood status | The EmojiGrid is administered immediately before and after viewing each laughter video on each day of the five-day intervention. Subjective mood status is assessed on day 1, 2, 3, 4, and 5 of the intervention both pre and post video viewing.
  Subjective mood status before and after each online video is viewed will be assessed using the EmojiGrid. The EmojiGrid is administered before and after viewing each video on each day of the five-day intervention (intervention group participants only).
  EmojiGrid has 17 emojis in total and is divided into four sets with five emojis each. In our study, set (A) was used with the question, "Using the emoji below, indicate how you feel right now." In addition, the researcher added a number to each emoji to help participants select the emoji that represented them at the time asked. The score ranges from 1-5, where higher numbers indicate happier mood states and lower numbers suggest lower mood, with 3 representing a neutral mood.

CONTACTS AND LOCATIONS:
Locations (1):
- Zayed University, Abu Dhabi, United Arab Emirates

IPD SHARING:
Plan to Share IPD: Undecided